CLINICAL TRIAL: NCT00110162
Title: A Collaborative Randomized Phase III Trial: The Timing of Intervention With Androgen Deprivation in Prostate Cancer Patients With Rising PSA
Brief Title: Androgen Deprivation Therapy in Treating Patients With Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: PMCC-VCOG-PR-0103; CDR0000413706 (Registry Identifier: PDQ (Physician Data Query)); PMCC-TROG-0306
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Orchiectomy

INTERVENTIONS:
Drug: antiandrogen therapy
Drug: releasing hormone agonist therapy
Procedure: orchiectomy

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Androgen deprivation therapy may stop the adrenal glands from making androgens.

PURPOSE: This randomized phase III trial is studying how well androgen deprivation therapy works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival (with acceptable morbidity) of patients with prostate cancer treated with delayed vs immediate androgen deprivation therapy (ADT).

Secondary

* Compare cancer-specific survival of patients treated with these regimens.
* Compare clinical progression in patients treated with these regimens.
* Compare time to first androgen independence in patients treated with these regimens.
* Compare complication rate incidence and timing (e.g., cord compression or pathological failure) in patients treated with these regimens.
* Compare treatment-related morbidity (including cognitive morbidity or osteoporosis) in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Determine prognostic factors for progression in patients treated with delayed ADT.

OUTLINE: This is a multicenter, randomized, controlled study. Patients in group 1 are stratified according to prior therapy (prostatectomy vs radiotherapy vs prostatectomy and radiotherapy), relapse-free interval (< 2 years vs ≥ 2 years), type of planned androgen deprivation therapy (ADT) (continuous vs intermittent), and participating center. Patients in group 2 are stratified according to type of planned ADT (continuous vs intermittent), disease type (localized vs metastatic), and participating center. Patients in both groups are randomized to 1 of 2 treatment arms.

* Arm I (delayed ADT): Beginning at least 2 years after study entry or after exhibiting evidence of significant disease progression*, patients receive either continuous ADT OR intermittent ADT comprising either bilateral orchiectomy OR luteinizing hormone-releasing hormone agonist with or without oral antiandrogen therapy.
* Arm II (immediate ADT): Beginning immediately after randomization, patients receive either continuous ADT OR intermittent ADT as in arm I.

NOTE: *Patients in group 1 begin delayed ADT at least 2 years after study entry unless 1 of the following clinical criteria is present: prostate-specific antigen (PSA) doubling time of < 12 months with PSA ≥ 10 ng/mL OR PSA doubling time of ≤ 6 months based on 3 consecutive measurements obtained ≥ 2 months apart OR development of metastases or symptoms. Patients in group 2 begin delayed ADT at least 2 years after study entry unless 1 of the following clinical criteria is present: development of symptoms OR PSA ≥ 60 ng/mL OR PSA doubling time of ≤ 6 months based on 3 consecutive measurements obtained ≥ 2 months apart.

After 9 months of ADT, all patients are assessed for response. Patients with PSA < 4 ng/mL may discontinue ADT. These patients are followed every 3 months. Treatment may be restarted when PSA is > 20 ng/mL OR PSA is > the PSA level at study entry OR at clinical progression.

Quality of life is assessed at baseline, every 6 months for 2 years, and then annually for 3 years.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then periodically thereafter at the discretion of the principal investigator.

PROJECTED ACCRUAL: A total of 300-2,000 patients will be accrued for this study within 2-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Prostate-specific antigen (PSA) relapse OR incurable disease diagnosed within the past 2 months AND meets criteria for either of the following groups:

  * Group 1

    * In PSA relapse after definitive radical treatment (prostatectomy or radiotherapy), as evidenced by 1 the following:

      * Post-prostatectomy PSA level ≥ 0.2 ng/mL
      * At least 3 rising PSA levels (post-radiotherapy) obtained ≥ 1 month apart, with the last PSA obtained within the past 2 months
    * No metastatic disease by bone scan or abdomino-pelvic CT scan
  * Group 2

    * Not suitable for radical treatment at primary diagnosis
    * Not planning to receive curative treatment
    * Localized or metastatic disease

      * No symptomatic disease requiring radiotherapy or immediate hormonal therapy
* No symptomatic disease requiring therapy

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* At least 5 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other significant comorbid condition that would limit life expectancy to < 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* At least 12 months since prior androgen deprivation therapy (ADT) administered in the neoadjuvant or concurrent (with radiotherapy) setting (group 1)
* No prior ADT (group 2)

Radiotherapy

* See Disease Characteristics
* See Endocrine therapy

Surgery

* See Disease Characteristics

Other

* No concurrent enrollment in TROG-96.01 or TROG-RADAR protocols

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2004-10; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Death from any cause at 8 years

SECONDARY OUTCOMES:
Cancer specific survival
Clinical progression
Time to first androgen independence
Complication rate incidence and timing (e.g., cord compression, pathological fracture)
Treatment-related morbidity (including cognitive, osteoporosis)
Prognostic factors for progression (delayed group)
EORTC Quality of life - general QLQC30 and prostate module for Quality of life annually for 5 years
CTC v3.0 Survival endpoints: actuarial analysis at eight years
Morbidity continuously

CONTACTS AND LOCATIONS:
Overall Officials: Gillian M. Duchesne, MD, FRCR, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (20):
- Australia (17):
  - Cancer Therapy Centre at Campbelltown Hospital, Campbelltown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Cancer Care Centre at Nepean Hospital, Kingswood, New South Wales
  - Cancer Therapy Centre at Liverpool Hospital, Liverpool, New South Wales
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - East Coast Cancer Centre, Tugun, Queensland
  - Urological Solutions, Ashford, South Australia
  - Repatriation General Hospital, Daws Park, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - West Gippsland Hospital, Warragul, Victoria
  - Christchurch Hospital, Christchurch
- New Zealand (3):
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North

REFERENCES:
- [Derived] Duchesne GM, Woo HH, King M, Bowe SJ, Stockler MR, Ames A, D'Este C, Frydenberg M, Loblaw A, Malone S, Millar J, Tai KH, Turner S. Health-related quality of life for immediate versus delayed androgen-deprivation therapy in patients with asymptomatic, non-curable prostate cancer (TROG 03.06 and VCOG PR 01-03 [TOAD]): a randomised, multicentre, non-blinded, phase 3 trial. Lancet Oncol. 2017 Sep;18(9):1192-1201. doi: 10.1016/S1470-2045(17)30426-6. Epub 2017 Jul 28. PMID 28760403
- [Derived] Duchesne GM, Woo HH, Bassett JK, Bowe SJ, D'Este C, Frydenberg M, King M, Ledwich L, Loblaw A, Malone S, Millar J, Milne R, Smith RG, Spry N, Stockler M, Syme RA, Tai KH, Turner S. Timing of androgen-deprivation therapy in patients with prostate cancer with a rising PSA (TROG 03.06 and VCOG PR 01-03 [TOAD]): a randomised, multicentre, non-blinded, phase 3 trial. Lancet Oncol. 2016 Jun;17(6):727-737. doi: 10.1016/S1470-2045(16)00107-8. Epub 2016 May 4. PMID 27155740